CLINICAL TRIAL: NCT02371421
Title: Genomic Guided Assessment of Drug Therapy Effectiveness in Managing Hmong Adults With Hyperuricemia or Gout.
Brief Title: Genetics of Hyperuricemia Therapy in Hmong
Acronym: GOUT-H
Status: Completed | Type: Observational
Sponsor: University of Minnesota (Other)
Responsible Party: Sponsor
Other Study IDs: 1408M53223
Record Dates: First submitted 2015-02-19; First posted 2015-02-25 (Estimated); Last update posted 2019-07-15 (Actual); Status verified 2019-07

CONDITIONS: Hyperuricemia, Gout
MeSH Terms: conditions — Hyperuricemia; Gout | interventions — Allopurinol

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Allopurinol: Participants with history of gout indicated by the use of allopurinol or participants who have high serum uric acid without contraindication to use allopurinol.
  Interventions: Drug: Allopurinol

INTERVENTIONS:
Drug: Allopurinol

SUMMARY:
To pursue this objective, we will be measuring uric acid at baseline and post 14 days of twice daily allopurinol therapy in 30 Hmong participants with documented gout or hyperuricemia and known genotype for key renal transporters of uric acid.

DETAILED DESCRIPTION:
Minnesota Hmong are a unique population of individuals of South East Asian descent who have been noted to have a higher prevalence of gout and gout related comorbidities compared to non-Hmong. Elevated levels of uric acid are thought to be at the root cause of gout. Elevated levels of serum uric acid can result from either overproduction and or under-excretion. Xanthine oxidase plays a key role in the breakdown of purines to form uric acid. Transporters in the kidney also play a key role in excretion and/or re-absorption of uric acid. The objective of this study is to explore whether genetic variations in renal transporters may influence the disposition of serum uric acid in response to a drug (allopurinol) as well as the disposition of its active metabolite (oxipurinol) which may also be a substrate for these same transporters responsible for uric acid disposition. Genetic variations unique to the Hmong population may explain their increased prevalence in gout and or perceived lack of responsiveness to the drug (allopurinol) used to treat the condition.

ELIGIBILITY:
Inclusion Criteria:

* Both parents are Hmong (self report)
* Self report history of gout, or
* History (within one year) of active use of xanthine oxidase inhibitors, or
* Evidence of serum uric acid ≥ 6mg/dL , or
* Serum uric acid < 6mg/dL with history of ≥ 2 gout episodes within the last 6 months
* Ability to provide informed consent for participation in the study
* Demonstrate understanding of the study procedures and ability to comply with the study drug for the entire length of the study
* Ability to obtain permission from treating clinician to allow stopping the drug for 10 days

Exclusion Criteria:

* Pregnant women or women of childbearing age sexually active and not using any contraception
* estimated creatinine clearance (eCrCl) <30ml/min
* Elevated liver enzymes (3 x upper normal limit of liver function tests (AST and ALT))
* Contraindication to receiving allopurinol
* Active participation in other clinical trial (or within 30 days)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Hmong (self-report) adulst with gout as evidenced by use of uric acid-reducing medication.
Sampling Method: Probability Sample
Enrollment: 80 (Actual)
Dates: Start 2014-06 (Actual); Primary Completion 2015-12 (Actual); Study Completion 2016-12 (Actual)

PRIMARY OUTCOMES:
Percent change from baseline in serum uric acid | 14 days
Steady state oxipurniol area under the serum concentration-time curve (AUC) | 14 days
  Differences in mean AUC across genotype groups

SECONDARY OUTCOMES:
Percent change from baseline in Uric Acid Fractional Excretion | 14 days
Percent change from baseline in Uric Acid Renal Clearance | 14 days

CONTACTS AND LOCATIONS:
Overall Officials: Robert J Straka, PharmD, Principal Investigator — University of Minnesota
Locations (1):
- University of Minnesota, Minneapolis, Minnesota, United States